CLINICAL TRIAL: NCT00002249
Title: A Double-Blind Study to Evaluate the Safety and Pharmacokinetics of L-Ofloxacin (RWJ 25213) in Subjects With HIV Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: R W Johnson Pharmaceutical Research Institute (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 105A/B; K90-086; K90-024
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1991-09

CONDITIONS: HIV Infections
Keywords: Anti-Infective Agents, Quinolone; Ofloxacin; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Levofloxacin

INTERVENTIONS:
Drug: Levofloxacin

SUMMARY:
To determine the safety and pharmacokinetics of L-ofloxacin (RWJ 25213) in patients with HIV infection.

ELIGIBILITY:
Inclusion Criteria

Patients must have the following:

HIV infection.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Active opportunistic infection or neoplasm.
* High likelihood of death during study.
* Significant ophthalmologic, renal, hepatic, cardiovascular, hematologic, neurologic, psychiatric,respiratory, or metabolic disease.
* Donation of > 1 unit blood or acute loss of blood within one month of study entry.

Patients with the following prior conditions are excluded:

* History of opportunistic infection.
* Previous allergic reaction to ciprofloxacin, norfloxacin, or any other quinolone.

Prior Medication:

Excluded:

Use of any investigational agent within 7 days of entry into study. Use of any medication within 3 days prior to entry (7 days for AZT). Alcohol or drug abuse.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- R W Johnson Pharmaceutical Research Institute, Raritan, New Jersey, United States

REFERENCES:
- [Background] Goodwin SD, Gallis HA, Chow AT, Wong FA, Flor SC, Bartlett JA. Pharmacokinetics and safety of levofloxacin in patients with human immunodeficiency virus infection. Antimicrob Agents Chemother. 1994 Apr;38(4):799-804. doi: 10.1128/AAC.38.4.799. PMID 8031049